CLINICAL TRIAL: NCT04701073
Title: Lumbar Belt Benefit Compared to the Usual Care in the Treatment of Non-specific Low Back Pain -an Interventional, Prospective, Multicenter, Randomized, Open and Controlled Study
Brief Title: Lumbar Belt Benefit Compared to the Usual Care in the Treatment of Non-specific Low Back Pain
Acronym: LOMBACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thuasne (Industry)
Collaborators: RCTs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EC33; 2020-003201-54 (Registry Identifier: IDRCB number. French competent authority : ANSM)
Record Dates: First submitted 2020-12-17; First posted 2021-01-08 (Actual); Last update posted 2024-09-05 (Actual); Status verified 2024-09

CONDITIONS: Low Back Pain
Keywords: Low back pain; Lumbar belt; Functional capacity; Medicoeconomic; Compliance
MeSH Terms: conditions — Low Back Pain; Patient Compliance

STUDY DESIGN:
Intervention Model Description: An interventional, prospective, multicenter, randomized, open and controlled study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group "usual care" (No Intervention): Promotion of physical activity and taking usual medicines for pain relief
- Intervention group : lumbar belt (Experimental): wearing the LombaStab belt during 3 months in addition to usual care (promotion of physical activity and taking usual medicines for pain relief).
  Interventions: Device: LombaStab belt

INTERVENTIONS:
Device: LombaStab belt — Instruction given to the patient will be to wear the LombaStab belt from 4 to 8 hours per days, over the whole duration of the study (12 weeks). The investigator will explain to the patient how to adjust it.
  The LombaStab belt will be equiped with thermosensor to evaluate the belt wearing time at the end of the study.
  Arms: Intervention group : lumbar belt

SUMMARY:
Lumbar belt benefit compared to the usual care in the treatment of non-specific low back pain -an interventional, prospective, multicenter, randomized, open and controlled.study

DETAILED DESCRIPTION:
This is a controlled study, with randomization of the patients, which aims at evaluating the benefit and interest of wearing a new generation lumbar belt, in patients suffering from non-specific low back pain. This trial is also designed to provide quality of life data and to assess the medico-economic interest of wearing such a lumbar belt.

This is an interventional study with low risks and constraints that does not deviate from the local standard of care for enrolled patients. No invasive examination or procedure is performed; as such, there will be no additional risks for participating patients.

203 patients will be followed during 12 weeks in up to 20 investigational sites Patients meeting all eligibility criteria will be included in the study and randomized into one of the two following groups on a 1: 1 ratio.

* Control group "usual care": promotion of physical activity and taking usual medicines for pain relief
* Intervention group: wearing the LombaStab belt in addition to usual care (promotion of physical activity and taking usual medicines for pain relief).

Three visits will be performed:

* Inclusion visit - baseline D0 - V0
* Follow-up visit at week 4 (+/- 5 days) - V1
* Follow-up visit at week 12 (+/- 5 days) - V2

At inclusion visit, after verification of the eligibility criteria, data regarding patients will be collected: demographic data, low back pain history, medical and surgical history, concomitant medications.

At each visit will be performed:

* physical examinations and score assessment by the investigator: ODI score, finger-to-floor distance test, Schober Mac Rae test
* medical interview with patient in order to collect the following information: description of pain, drug consumption, duration of sick leave and resumption of activity at work, use of medical resources (consultations and complementary).
* reporting of all AEs and device deficiencies

Patients will be asked to complete on-line questionnaires, following visits and each week.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged from 18 to 55 years old
* Patient suffering from non-specific low back pain with current episode has progressed for 1 to 6 months
* At least one lumbar mean pain at rest or at effort of the last 72 hours collected on inclusion ≥ 40/100 on an NRS scale.
* Ability of the patient or legally authorized representative to provide a signed and dated i informed consent form before any procedure or data collection.
* Patient covered by the French Social security system.

Exclusion Criteria:

* Patient wearing a lumbar belt the day of the inclusion visit
* Patient who has had surgical intervention on dorso-lumbar spine or lower limb the past 5 years or who has planned surgery during the study
* MODIC diagnosis (disc degeneration) known or confirmed by MRI
* On sick leave for more than 3 consecutive months due to low back pain at the time of inclusion
* Low back pain related to an accident at work
* Low back pain due to secondary origin: tumor, inflammatory, infectious cause, related to a fracture or a vertebral compression
* Patient with fibromyalgia
* Patient with lumbar radicular syndrome (radicular conflict like disc herniation, spinal stenosis...)
* Pregnant woman or trying to become pregnant during the study
* Patient with confirmed depression
* Patient with cognitive or mental disorders
* Morphology with measurements not allowing to match with the sizes of belts available
* Patient presenting chronic pathology with disabling functional consequences
* Patient who received an infiltration less than one month before inclusion visit or planned during the study
* Patient with known allergy to any of the materials (see product composition in the Description section of user instruction)
* Patient with contraindicated to belt wearing: hiatus hernia, deficient respiratory functions
* Anticipated poor compliance of subject with study procedures
* Current participation in an interventional investigation drug or device treatment study with an impact on evaluation criteria

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 168 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Change from baseline ODI score (Oswestry Disability Index) at 12 weeks | Week: 0 and 12
  The functional capacity is measured by ODI score.The ODI questionnaire consists in 10 questions and 6 answers modalities.The ODI score results are expressed in percentage.The higher the percentage is, the more the functional capacity is impaired.

SECONDARY OUTCOMES:
Evolution of functional capacity | Week: 0 and 4
  The functional capacity is measured by ODI score.The ODI questionnaire consists in 10 questions and 6 answers modalities.The ODI score results are expressed in percentage.The higher the percentage is, the more the functional capacity is impaired.
Evolution of pain level | Week: 0, 4 and 12
  Pain level is measured by NRS scale completed by the patient : minimum, maximum, mean at effort and at rest : 0 corresponds to no pain (better outcome) and 10 to maximum pain (worst outcome)
Evolution of pain characteristics | Week: 0, 4 and 12
  Characteristics of pain are evaluated by specific questions regarding the description of pain
Evolution of Quality of Life | Week: 0 and 12
  Quality of life is measured by the EQ5D questionnaire completed by the patient. The EQ-5D questionnaire has two components: health state description and evaluation.
  In the description part, health status is measured in terms of five dimensions (5D); mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Mobility dimension asks about the person's walking ability. Self-care dimension asks about the ability to wash or dress by oneself, and usual activities dimension measures performance in "work, study, housework, family or leisure activities". In pain/discomfort dimension, it asks how much pain or discomfort they have, and in anxiety/depression dimension, it asks how anxious or depressed they are. The respondents self-rate their level of severity for each dimension using five-level (EQ-5D-5L) scale.
  In the evaluation part, the respondents evaluate their overall health status using the visual analogue scale (EQ-VAS).
Assessment of doctors' opinion on improving the patient's health condition caused by low back pain and severity | Week 0, 4 and 12
  Improvement and severity are measured by the CGI-I and CGI-S questionnaires respectively.
  Doctors' opinion on the change of patient's health condition due to low back pain is measured by the Clinical Global Impression - Improvement questionnaire. The scale has 7 levels of answer from "very strongly improved" which is the better outcome (= 1 point) to "very strongly aggravated" which is the worst outcome (= 7 points) .Intermediate levels are: " Significantly improved "(= 2 points) ; " Slightly improved " (= 3 points) ; " No improvement " (=4 points) ; " Slightly worsen " (=5 points) ; " Seriously worsen" ( = 6 points).
  The highest score corresponds to the most impairment in quality of life.
Assessment of patient's opinion on Global Impression of Change about his general condition | Week: 4 and 12
  Improvement is measured by the PGI-C questionnaire. Patient's opinion on Global Impression of Change about her general condition is measured by the modified PGI-C questionnaire (Patient's opinion on Global Impression of Change). The scale has 7 levels from "no change or condition has got worsed"(worse outcome) to "a great deal better, and a considerable improvement that has made all the difference ( better outcome)". Intermediate levels are: "almost the same, hardly any change at all"; "a little better, but no noticeable change", "somewhat better, but the change has not made any real difference"; "moderately better, and a slight but noticeable change"; "better, and a definite improvement that has made a real and worthwhile difference.
Evolution of spinal mobility vie Finger to floor distance test | Week: 0, 4 and 12
  Spinal mobility is measured by finger-to-floor distance test. The subject stands erect on a platform 20-cm high He's asked to bend forward as far as possible, while maintaining the knees, arms, and fingers fully extended. The vertical distance between the tip of the middle finger and the platform is measured with a suppletape measure in centimeters. The vertical distance between the platform and tip of the middle finger is positive when the subject do not reach the platform and negative when he can go further.
Evolution of spinal mobility via Schober Mac Rae test | Week: 0, 4 and 12
  Spinal mobility is measured by Schober Mac Rae test. The Patient is standing, examiner marks both posterior superior iliac spine and then draws a horizontal line at the centre of both marks. A second line is marked 5 cm below the first line.
  A third line is marked 10 cm above the first line. Patient is then instructed to flex forward as if attempting to touch his/her toes, examiner remeasures distance between the top and bottom line.
Evolution of physical activity | Week: 0, 4 and 12
  Physical activity is measured by IPAQ questionnaire completed by the patient The IPAQ questionnaire measures the time associated to intensive activity, moderate activity, walking and sitting in the last week.
Evolution of drug consumption | Week: 0, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11 and 12
  Drug consumption (analgesics, anti-inflammatories, etc), is recorded by the patient each week in ePRO (name of the drug, frequency of taking the medication)
Medical and paramedical consultations | Week: 0, 4 and 12
  Number of consultations (physiotherapy / doctors / osteopathy…) or hospitalization and complementary examinations carried out are measured by patient's interview
Duration of Sick leave | Week: 0, 4 and 12
  Global duration of sick leave (number of days, Saturday and Sunday included) is measured by patient's interview
Assessment of tolerance | Week: 4 and 12
  Tolerance is measured by adverse events reported. Number and type of serious and non-serious Adverse Device Effects (ADE) are reported..
Assessment of time of belt's wearing | through study completion, an average of 12 weeks
  Compliance is measured by a thermosensor specific device fixed to the belt
Assessment of patient's satisfaction about the lumbar belt comfort and design | Week 12
  Satisfaction is measured by a specific questionnaire completed by the patient. Questions are about comfort, easy to use, performance on pain, aesthetic...

CONTACTS AND LOCATIONS:
Overall Officials: Laurent GRANGE, MD, PH, Principal Investigator — CHU de Grenoble Alpes
Locations (3):
- France (3):
  - CHU Grenoble Alpes, Grenoble
  - Hôpital Cochin, Paris
  - CHU de St Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No